# Strengthening Healthy Relationships Among Apsaalooke Youth NCT05734014 Unique Protocol Id 4W8808 April 29, 2024

# **Study Protocol**

<u>Study Purpose</u>: The purpose of this study is to conduct a feasibility and acceptability of a pilot intervention to promote relationality among Apsáalooke youth. This formative study is grounded in community-based participatory efforts to build locally relevant educational programming for youth and support the development of future evidence-based programming for youth.

# Participants and Inclusion Citeria:

Participants in this study consisted of youth maximum age of 13 who are enrolled in 5<sup>th</sup>-6<sup>th</sup> grade at the time of the study. Eligibility criteria included youth that live on or near the Crow Reservation in Montana and have parental or guardian consent to participate. Recruitment efforts were conducted in partnership with local schools, educational liaisons, and community champions. Information about the program was shared through school announcements, flyers sent home with students and presentations during school-based and community events. Interested families received informational packets and consent forums outlining the purpose, procedures and voluntary nature of participants. Informed consent was also obtained from parents and assent from each youth participant. The recruitment spanned from May 2024 through June 2024. A total of 10 participants were recruited and enrolled in the study.

### **Data Collection Methods**

Data for this feasibility study consisted of process evaluation data and qualitative, art-based reflections. The primary data collected included recruitment and retention metrics: Researchers tracked the number of students recruited, consented, and retained during the program. Session Observations: Trained facilitators and researchers documented implementation fidelity, student engagement, and logistical issues during sessions. Observational field notes were compiled systematically and informed the overall assessment of feasibility.

Arts-based qualitative reflections. At the conclusion of each session, students participated in a reflective activity using paper and markers to draw or write about their experiences. Prompts included: "What did you like best today?" "What did you learn?" "What would you like to share with your family?" The creative responses provided insight into the youth's internalization of key messages and their personal engagement with the content. Following the acidity, students voluntarily shared their drawing and narratives with the group. Researchers took detailed notes during these sharing moments to record accurate explanations.

### Data Analysis

At thematic approach was used to analyze the qualitative data from the arts-based discussion. Drawings and reflections were reviewed coded and categorized to identify salient themes across participant responses. Themes were co-analyzed by research team member to ensure relevance and interpretive validity. Observational data were reviewed alongside participant responses to assess consistency between program delivery and participant experience. The study was conducted in alignment with community based participatory research principles.